CLINICAL TRIAL: NCT05363735
Title: Ultrasound Elastography Application in the Assessment of Cesarean Section Scar Defect.
Brief Title: Ultrasound Elastography Application in Cesarean Section Scar Defect
Status: Withdrawn | Type: Observational
Why Stopped: Device can't meet the requirements
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-21-015
Record Dates: First submitted 2022-03-19; First posted 2022-05-06 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2022-05

CONDITIONS: Cesarean Section; Dehiscence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasound Elastography: Patients will be examined by ultrasound elastography.
  Interventions: Other: Ultrasound Elastography

INTERVENTIONS:
Other: Ultrasound Elastography — Patients will be examined by ultrasound elastography.

SUMMARY:
Cesarean Section Scar Defect(CSD) is one of the complications after cesarean section. CSD will cause many long term complications, such as abnormal uterine bleeding, infertility, uterine scar pregnancy and uterine rupture. Transvaginal ultrasound was used to detect uterine scar defects commonly. Ultrasound elastography is a modern imaging technique that has developed rapidly in recent years. Thus, this study intend to investigate the application of Ultrasound Elastography in Cesarean Section Scar Defect.

ELIGIBILITY:
Inclusion Criteria:

* Clearly diagnosed with CSD
* No serious medical problems (important viscera function in the normal range). uterine fibroids no more than 5cm
* Sign the informed consent.

Exclusion Criteria:

* Indefinite diagnosis.
* Malignant tumors.
* With severe medical problems (severe liver disease, kidney disease, respiratory diseases, heart disease or uncontrolled diabetes, epilepsy, etc., dysfunction of important organs).
* Pregnant.
* Mental diseases.
* Unwilling to comply with the research plan.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: women who were diagnosed with CSD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
thickness of the remaining muscular layer | 4 weeks before vaginal repair of CSD
  The thickness of the remaining muscular layer is measured by ultrasound
thickness of the remaining muscular layer | 12 weeks after vaginal repair of CSD
  The thickness of the remaining muscular layer is measured by ultrasound
strain ratio (SR) | 4 weeks before vaginal repair of CSD
  the ratio of mean strain in the lesion to the adjacent background tissue
strain ratio (SR) | 12 weeks after vaginal repair of CSD
  the ratio of mean strain in the lesion to the adjacent background tissue

CONTACTS AND LOCATIONS:
Overall Officials: Wang Xipeng, Dr, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided